CLINICAL TRIAL: NCT01130064
Title: A Multi-center, Randomized, Double Blind, Placebo-controlled, 'add-on' Study to Investigate the Efficacy and Safety of 24 Weeks Intravenous Treatment With QAX576 in Patients (≥18-75 Years) With Persistent Asthma Not Adequately Controlled With Inhaled Corticosteroids and Long Acting β2-agonists
Brief Title: Efficacy of QAX576 in Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAX576A2207; 2009-011590-32 (EudraCT Number)
Record Dates: First submitted 2010-05-24; First posted 2010-05-25 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2017-02

CONDITIONS: Asthma
Keywords: Asthma; QAX576
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- QAX576 (Experimental): QAX576
  Interventions: Biological: QAX576
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: QAX576 — every 3 weeks via intravenous infusion
  Arms: QAX576
Drug: Placebo — every 3 weeks via intravenous infusion
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the efficacy of 24 weeks intravenous treatment with QAX576 in patients with persistent asthma not adequately controlled with inhaled corticosteroids and long acting beta2-agonists.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* Female patients must be surgically sterilized or postmenopausal
* Male patients must use two forms of contraception
* Body mass index must be between 18 and 39 kg/m2
* Diagnosis of asthma for at least one year, which is not adequately controlled by inhaled corticosteroids and long acting beta-2 agonists

Exclusion Criteria:

* Smoking history >10 pack-years
* Patients with a diagnosis of chronic obstructive pulmonary disease (COPD)
* Patients who have experienced a severe asthma attack/exacerbation requiring systemic corticosteroids or an increase in maintenance doses, within 6 weeks of screening
* Patients who have had a respiratory tract infection within 6 weeks prior to screening
* History of schistosomiasis, within 6 months of screening, or traveling to a country endemic with schistosomiasis within 6 months of completing the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2010-05; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Asthma Control Questionnaire | 24 weeks

SECONDARY OUTCOMES:
Incidence rate of clinically significant asthma exacerbations | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (44):
- United States (10):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Huntington Beach, California
  - Novartis Investigative Site, Owensboro, Kentucky
  - Novartis Investigative Site, Wheaton, Maryland
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Marion, Ohio
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Summerville, South Carolina
- Argentina (5):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Mendoza
  - Novartis Investigative Site, Santa Fe
- Belgium (6):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Eupen
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Laken
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
- Czechia (4):
  - Novartis Investigative Site, Rokycany, Czech Republic
  - Novartis Investigative Site, Strakonice, Czech Republic
  - Novartis Investigative Site, Teplice, CZE
  - Novartis Investigative Site, Tábor
- Germany (7):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Großhansdorf
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Rüdersdorf
- Poland (5):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Poznan
- Russia (7):
  - Novartis Investigative Site, Kazan', Tatarstan Republic
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Samara
  - Novartis Investigative Site, Yaroslavl

REFERENCES:
- See also: Results for CQAX576A2207 from Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=8063